CLINICAL TRIAL: NCT01991548
Title: A User Evaluation of the MiniMed® 640G Insulin Pump and Guardian® Link Transmitter
Brief Title: User Evaluation of the MiniMed 640G Insulin Pump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP284
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2016-03

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Diabetic participants with study devices (Other)
  Interventions: Device: MiniMed® 640G Insulin Pump and Guardian® Link Transmitter

INTERVENTIONS:
Device: MiniMed® 640G Insulin Pump and Guardian® Link Transmitter

SUMMARY:
This four center international study will include two United Kingdom National Health Service centers, and two centers in Melbourne, Australia. The objective of the study is to evaluate subject acceptance of a new insulin pump and transmitter together with the accompanying training materials. Descriptive data from participant questionnaires and device uploads will be evaluated.

Pediatric subjects between the ages of 7 - 18 years and adults from the age of 19 years of age upwards, who currently use an insulin pump in the management of their type 1 or type 2 diabetes, will be invited to participate. Each subject will be trained on the study device and then use it for approximately four weeks. During this time there will be three in-clinic visits and four follow-up phone calls, scheduled at the subjects' convenience. At the end of this period, they will revert back to their original insulin pump and complete a questionnaire on the study pump training materials, features and usability.

ELIGIBILITY:
Criteria for Inclusion: A subject is eligible for the user evaluation study if all of the following criteria are met:

1. Subject is 7 years or older at time of screening
2. Subject is current insulin pump user for at least 3 months
3. Subject has the following CGM experience as determined by the Investigator:

   * Has experience and is able to insert/change sensor by herself/himself and
   * Has experience and can recharge the transmitter and
   * Has experience and can read sensor data in real-time on her/his pump screen
4. Subject/legal representative has signed a Patient Informed Consent and is willing to comply with the study procedures;
5. Subject is willing to complete study questionnaires throughout the study
6. Must have the following clinical diagnosis:

1. Type 1 diabetes, for a minimum of 6 months prior to enrollment

Criteria for Exclusion: A subject is excluded from the user evaluation if any of the following criteria are met:

1. Female subject has a positive urine pregnancy screening test.
2. Female subject who plans to become pregnant during the course of study. If a woman becomes pregnant during participation, she will be withdrawn
3. Subject has any condition that, in the opinion of the Investigator or qualified Investigational Centre staff, may preclude him/her from participating in the study and completing study related procedures.
4. Subject has impaired vision or hearing problems that could compromise the handling of the device as determined by Investigator or qualified Investigational Centre staff
5. Subject is unable to tolerate tape adhesive in the area of sensor placement
6. Subject has any unresolved adverse skin condition in the area of sensor placement (e.g. psoriasis, rash, Staphylococcus infection)
7. Subject has travel plans which would make it difficult for the subject to attend on-site study visits as scheduled
8. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks (CEP267 User Evaluation is not included in this exclusion criteria).

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (2):
  - St Vincent Hospital and The University of Melbourne, Fitzroy
  - The Royal Melbourne Hospital, Patkville
- United Kingdom (2):
  - University College Hospital, London
  - King's College London, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Dependent Diabetics: Subjects currently using an insulin pump transferred to use the Medtronic MiniMed 640G insulin pump and Guardian Link transmitter.
Period: Overall Study
Arm/Group | Insulin Dependent Diabetics
Started | 40
Completed | 39
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Insulin Dependent Diabetics: individuals with insulin dependant diabetes using the 640G insulin pump for insulin infusion and continuous glucose monitoring
Arm/Group | Insulin Dependent Diabetics
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (17.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: User Acceptance of the New MiniMed 640G Insulin Pump and Guardian Link Transmitter
Description: Descriptive summary will be used to characterize the results of the study questionnaires. The questionnaire will use a Likert scale (rating of 1 to 7) to assess subject acceptance of the MiniMed 640G, Guardian Link Transmitter, and the training materials. A response of 4 or greater will be considered positive on a Likert scale for training materials and product acceptance.
Time Frame: Four weeks of pump wear
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Overall: Descriptive summary will be used to characterize the results of the study questionnaires. The questionnaire will use a Likert scale (rating of 1 to 7) to assess overall subject acceptance of the MiniMed 640G and Guardian Link Transmitter. A response of 4 or greater on the Likert scale will be considered positive and indicate and product acceptance.
Arm/Group | Overall
Number analyzed (Participants) | 50
units on a scale | 6.02 (1.13)

ADVERSE EVENTS:
Time Frame: October 24, 2014 through November 12, 2014
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 4/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=40)
Dermatitis contact (General disorders) | 2 (2) — Allergic reaction to tape
Nasopharyngitis (Infections and infestations) | 1 (1) — Common cold
Urinary tract infection (Infections and infestations) | 1 (1) — Urinary tract infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No